CLINICAL TRIAL: NCT04048447
Title: Endoscopic Characterization of Colorectal Neoplasia With the Different Published Classifications: a Prospective Comparative Study Involving Gastroenterologists From Trainees to Experts.
Brief Title: Endoscopic Characterization of Colorectal Neoplasia With the Different Published Classifications
Status: Completed | Type: Observational
Sponsor: Hôpital Edouard Herriot (Other)
Responsible Party: Principal Investigator, Jean Christophe Saurin, Professor, Hôpital Edouard Herriot
Other Study IDs: SFED PROTOCOL
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Colorectal Neoplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endoscopic characterization is now essential in front of a colorectal lesion to predict its histology and choose the best therapeutic strategy. Different classifications have been proposed to predict histology depending on the endoscopic aspect. Thus, the aspect of the shape of the lesion is described in the Paris classification, the aspect of the mucosal pattern in Kudo's classification and the vascular pattern in Sano's one. Recently, classifications combining several color and mucosal and vascular pattern criteria have been described as the NICE classification or even more recently the Japanese JNET classification. However, although the interest in combining the Paris, Sano and Kudo criteria has recently shown its interest, there was not yet an overall classification covering all the published criteria. We have created a synthetic classification called CONECCT grouping the different criteria for an initial educational purpose. We have demonstrated that this tool allows interns and gastroenterologists to progress in the histological prediction of colorectal lesions presented in the form of photo files. Nevertheless, comparative data of the performances of those different classifications to predict the histology and the concordance intra and inter-observer have never been published. To validate this CONECCT classification, we created this comparative study evaluating the endoscopic characterization performances of these different classifications in terms of histological prediction and intra- and interobserver concordance in a group of gastroenterologists with varying levels of expertise in front of colorectal lesions presented in the form of photographic records.

ELIGIBILITY:
Inclusion Criteria:

* The participants were gastroenterologist doctors (experts, general or internal).
* Lesions presented were resected endoscopically after completion of a picture file.
* Pathology available for presented lesions.
* Participants signed informed consent and voluntarily participated in the characterization of these 206 lesions.

Exclusion Criteria:

* None

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Colic Neoplasia Patients
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the interobserver Concordance of the CONECCT classification compared to the 6 other existing ones | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Edouard Herriot Hospital, Lyon, Auvergne-Rhône-Alpes, France